CLINICAL TRIAL: NCT07154784
Title: Long-term Efficacy and Safety of Fecal Microbiota Transplantation in Patients With Ulcerative Colitis
Status: Enrolling by invitation | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Seoul National University Bundang Hospital (Other); Inha University Hospital (Other); Seoul National University Boramae Hospital (Other)
Responsible Party: Principal Investigator, KwangWoo Kim, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-0314
Record Dates: First submitted 2025-07-08; First posted 2025-09-04 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-08

CONDITIONS: Ulcerative Colitis; Fecal Microbiota Transplantation
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ulcerative colitis patient (Experimental): This was a multicenter, prospective study that enrolled patients diagnosed with ulcerative colitis who were aged between 10 and 80 years and had been receiving treatment for at least 3 months. Eligible participants were required to meet all of the following inclusion criteria:
  1. age between 10 and 80 years;
  2. a disease duration of ulcerative colitis of at least 3 months;
  3. mild to moderate disease activity, defined by a Mayo score of 4-10 or a partial Mayo score of 2-7;
  4. endoscopic evidence of rectal involvement extending ≥5 cm; and
  5. willingness to provide written informed consent for participation in the study.
  Interventions: Biological: Fecal microbiota transplantation (FMT)

INTERVENTIONS:
Biological: Fecal microbiota transplantation (FMT) — Fecal microbiota transplantation (FMT) will be performed at weeks 0 and 4 of study enrollment by administering approximately 250-300 cc of a multi-donor fecal suspension into the colon via sigmoidoscopy, colonoscopy, or by oral administration of an equivalent amount (4 capsules).

SUMMARY:
This study aims to perform fecal microbiota transplantation (FMT) and analyze its effects in selected patients aged between 10 and 80 years who have been diagnosed with ulcerative colitis and have been receiving treatment for more than three months at Seoul National University Hospital, Seoul National University Boramae Medical Center, and Seoul National University Bundang Hospital. Through this analysis, the study seeks to identify the long-term efficacy of FMT as a treatment for ulcerative colitis, evaluate the safety of the procedure, and establish a foundation for personalized FMT based on gut microbiota analysis.

DETAILED DESCRIPTION:
The pathogenesis of inflammatory bowel disease (IBD) is thought to result from a complex interplay of genetic predisposition, environmental factors such as diet and gut microbiota, and immunological mechanisms. Among these, increasing attention has been given to the role of the gut microbiota, which resides on the intestinal mucosal surface and plays a key role in regulating host immune responses. Emerging evidence suggests that alterations in gut microbiota, as well as viruses that influence microbial composition, are closely associated with IBD.

In 2013, a landmark study published in the New England Journal of Medicine demonstrated that fecal microbiota transplantation (FMT)-a procedure in which processed stool from a healthy donor is delivered into a patient's colon via colonoscopy-significantly reduced the recurrence of antibiotic-associated Clostridioides difficile infection. Since then, FMT has been actively studied, particularly for its therapeutic potential in ulcerative colitis, a subtype of IBD.

Randomized controlled trials have investigated various methods of FMT delivery in ulcerative colitis, including colonoscopy, sigmoidoscopy, and oral capsules. No significant differences in efficacy have been reported between endoscopic and oral routes. In a domestic study on multidrug-resistant organisms, oral capsules showed promising outcomes in restoring microbial balance when compared with endoscopy and nasogastric tube administration.

While FMT delivery methods in Western countries are evolving from inpatient colonoscopic administration to outpatient enema or capsule-based regimens, South Korea currently lacks clinical research infrastructure for FMT beyond case reports. Although a few cases of FMT in IBD patients have been documented, no center has conducted formal clinical trials.

Therefore, this study aims to evaluate the clinical efficacy and underlying mechanisms of FMT in Korean patients with IBD, especially those with ulcerative colitis. Through this investigation, we seek to clarify the long-term therapeutic potential and safety of fecal microbiota transplantation in this population.

ELIGIBILITY:
Inclusion Criteria:

* Age between 10 and 80 years
* History of ulcerative colitis for at least 3 months
* Mild to moderate ulcerative colitis with a Mayo score of 4-10 or a partial Mayo score of 2-7
* Endoscopic evidence of rectal involvement extending at least 5 cm
* Willingness to provide written informed consent for participation in this clinical trial

Exclusion Criteria:

* Hospitalization due to acute severe ulcerative colitis (Mayo score 11-12)
* Neutropenia (absolute neutrophil count < 500)
* Pregnancy
* Infectious colitis not caused by Clostridioides difficile
* History of colectomy (excluding appendectomy)
* History of antibiotic use within the past 2 weeks
* Use of corticosteroids > 20 mg within the past 4 weeks
* Current or planned use of biologics (e.g., anti-TNF-α antibodies, anti-α4β7 integrin monoclonal antibodies, JAK inhibitors, anti-IL-12/IL-23 antibodies)
* Major food allergy
* Indeterminate colitis
* Comorbid chronic diseases such as chronic liver disease, heart failure, or chronic obstructive pulmonary disease (COPD)
* Refusal to participate in the study
* Any other condition deemed inappropriate for study participation by the investigator

Ages: 10 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-07-19 (Actual); Primary Completion 2023-07-19 (Actual); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Co-primary outcome | The disease status will be evaluated at week 12 as the final assessment. Long-term efficacy and safety will also be analyzed at week 48(e.g., History of hospitalization, mortality, occurrence of malignant tumors, and adverse events[Safety]).
  1. Steroid-free Clinical Response at Week 12 Mayo score ≥3 and ≥30% ↓ from baseline, with rectal bleeding subscore ↓ ≥1 or ≤1, without steroid use.
     Unit: Participants
  2. Steroid-free Clinical Remission at Week 12 Mayo score ≤2 and no subscore >1, without steroid use. Unit: Participants

SECONDARY OUTCOMES:
Co-secondary outcome | The disease status will be evaluated at week 12 as the final assessment. Long-term efficacy and safety will also be analyzed at week 48(e.g., History of hospitalization, mortality, occurrence of malignant tumors, and adverse events[Safety]).
  1.Clinical Response at Week 12 and 48 Mayo ≥3 and ≥30%↓, rectal bleeding subscore ↓≥1 or ≤1. Unit: Participants
Co-secondary outcome | The disease status will be evaluated at week 12 as the final assessment. Long-term efficacy and safety will also be analyzed at week 48(e.g., History of hospitalization, mortality, occurrence of malignant tumors, and adverse events[Safety]).
  2.Clinical Remission at Week 12 and 48 Mayo ≤2 and all subscores ≤1. Unit: Participants
Co-secondary outcome | The disease status will be evaluated at week 12 as the final assessment. Long-term efficacy and safety will also be analyzed at week 48(e.g., History of hospitalization, mortality, occurrence of malignant tumors, and adverse events[Safety]).
  3.Endoscopic Response at Week 12 and 48 Mayo endoscopic subscore ↓≥1 from baseline. Unit: Participants
Co-secondary outcome | The disease status will be evaluated at week 12 as the final assessment. Long-term efficacy and safety will also be analyzed at week 48(e.g., History of hospitalization, mortality, occurrence of malignant tumors, and adverse events[Safety]).
  4.Endoscopic Remission at Week 12 and 48 Mayo endoscopic subscore = 0. Unit: Participants
Co-secondary outcome | The disease status will be evaluated at week 12 as the final assessment. Long-term efficacy and safety will also be analyzed at week 48(e.g., History of hospitalization, mortality, occurrence of malignant tumors, and adverse events[Safety]).
  5.CRP Change at Week 12 and 48 Change in serum CRP from baseline. Unit: mg/dL
Co-secondary outcome | The disease status will be evaluated at week 12 as the final assessment. Long-term efficacy and safety will also be analyzed at week 48(e.g., History of hospitalization, mortality, occurrence of malignant tumors, and adverse events[Safety]).
  6.ESR Change at Week 12 and 48 Change in ESR from baseline. Unit: mm/hr
Co-secondary outcome | The disease status will be evaluated at week 12 as the final assessment. Long-term efficacy and safety will also be analyzed at week 48(e.g., History of hospitalization, mortality, occurrence of malignant tumors, and adverse events[Safety]).
  7.Fecal Calprotectin Change at Week 12 and 48 Change from baseline. Unit: mg/kg
Co-secondary outcome | The disease status will be evaluated at week 12 as the final assessment. Long-term efficacy and safety will also be analyzed at week 48(e.g., History of hospitalization, mortality, occurrence of malignant tumors, and adverse events[Safety]).
  8.Microbiome Change at Week 12 and 48 Change in % relative abundance via 16S rRNA or shotgun. Unit: % relative abundance
Co-secondary outcome | The disease status will be evaluated at week 12 as the final assessment. Long-term efficacy and safety will also be analyzed at week 48(e.g., History of hospitalization, mortality, occurrence of malignant tumors, and adverse events[Safety]).
  9.Cytokine Change at Week 12 and 48 Change in mucosal cytokine levels from baseline. Unit: pg/mL
Co-secondary outcome | The disease status will be evaluated at week 12 as the final assessment. Long-term efficacy and safety will also be analyzed at week 48(e.g., History of hospitalization, mortality, occurrence of malignant tumors, and adverse events[Safety]).
  10.Single-cell RNA Expression Change at Week 12 and 48 Change in gene expression from serum (scRNA-seq). Unit: Fold change

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul Metropolitan Government Seoul National University Boramae Medical Center, Seoul National University College of Medicine, Seoul, Dongjak-gu, South Korea